CLINICAL TRIAL: NCT02370056
Title: Comparative Assessment of Three-dimensional vs. Conventional Laparoscopy in a Total Colectomy Model for Ulcerative Colitis
Brief Title: Evaluation of 3D Visualization for Total Colectomy
Acronym: 3Dvs2DforUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Emre Gorgun, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCFJJN4
Record Dates: First submitted 2015-02-09; First posted 2015-02-24 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3D Visualization (Experimental): 3-dimensional visualization: In this group, total laparoscopic abdominal colectomy will be performed for patients diagnosed with ulcerative colitis by using 3D Laparoscopic Surgical Video System.
  This group will be consisted of 27 patients, 9 colectomies performed by 3 surgeons.Effect of using 3D Laparoscopic Surgical Video System on operative outcomes will be evaluated.
  Interventions: Diagnostic Test: 3-dimensional visualization
- 2D Visualization (Active Comparator): 2-dimensional visualization: In this group, total laparoscopic abdominal colectomy will be performed for patients diagnosed with ulcerative colitis by using conventional Laparoscopic Surgical Video System.
  This group will be consisted of 27 patients, 9 colectomies performed by 3 surgeons and outcomes will be evaluated.
  Interventions: Diagnostic Test: 2-dimensional visualization

INTERVENTIONS:
Diagnostic Test: 3-dimensional visualization — Subjects are receiving Standard of Care Colectomy for Ulcerative Colitis visualized in 3D mode
  Arms: 3D Visualization
Diagnostic Test: 2-dimensional visualization — Subjects are receiving Standard of Care Colectomy for Ulcerative Colitis visualized in 2D mode
  Arms: 2D Visualization

SUMMARY:
The anticipated advantages of 3D laparoscopic visualization for the surgeon are greater accuracy and speed in manual skills, translating to decreased operative time, reduced learning curve, and superior safety.We aimed to determine the feasibility of the laparoscopic approach using 3D visualization in the surgical treatment of ulcerative colitis

DETAILED DESCRIPTION:
Three-dimensional (3D) visualization technology for laparoscopy has been proposed, since the early 1990's, as a method to facilitate laparoscopic performance. However, early 3D laparoscopic technology was limited in terms of image quality, so that its use had not been implemented. The latest technical developments ensure high-definition 3D visualization with the same quality that current two-dimensional (2D) systems provide.

The anticipated advantages of 3D laparoscopic visualization for the surgeon are greater accuracy and speed in manual skills, translating to decreased operative time, reduced learning curve, and superior safety . It was reported that, 3D laparoscopic visualization offers significant advantages in enhancing laparoscopic performance, even in novice surgeons, comparing to the 2D systems . We hypothesize that 3D visualization may allow surgeons to reduce the overall operating time with a rate of 10% with comparable perioperative and postoperative outcomes. The primary endpoint of this study is to determine the feasibility of the laparoscopic approach using 3D visualization in the surgical treatment of ulcerative colitis. Secondary endpoints are to determine whether 3D visualization confers benefits such as reduced operating time and intra-operative complications with comparable postoperative outcomes.

Device Description: The EXERA III Universal Platform will be used in this study, in conjunction with the ENDOEYE FLEX 3D. The ENDOEYE FLEX 3D can also be used in 2D mode, by utilizing a programmed button on the handle of the scope, or by using the 2D/3D button on the 3D Visualization Unit. The articulating tip of the ENDOEYE FLEX allows for the scope to be used in both single-site and multi-port procedures, providing critical views and allowing a bird's eye view so that the scope is out of the way of other instruments (while still capturing the image at the surgical site). All equipment used in this trial has been cleared under 510(k) approval by the FDA, and has been on the market in the US since April 2013.

The Olympus HD 3D Laparoscopic Surgical Video System consists of the following components:

* CV-190 Processor
* CLV-190 Light Source
* 3DV-190 3D Visualization Unit
* LMD-2451MT/3G4 Sony 24" 3D Monitor
* IMH-20 Image Capture System
* UHI-4 Insufflator
* K10021611 Cart
* OL-0015-08 Tall Rollstand
* LTF-190-10-3D ENDOEYE FLEX 3D Videoscope
* 3D glasses (regular and clip-on styles)

Study Size:Mean operating time for laparoscopic subtotal colectomy for medically refractory UC was reported longer with a comparison to open surgery in the recently published studies.

Therefore the effort to decrease operating time in laparoscopic colectomy has gained importance. We assumed that, in order to be able to determine a 10% reduction in mean operating time, each group should include 27 patients (80% power and 5% significance).

Patients who will undergo laparoscopic total abdominal colectomy (TAC) for UC will be included in the study. All subjects will be randomized into two groups: 3D laparoscopy, and 2D laparoscopy. Three staff surgeons (EG, HK, FR) at the department of colorectal surgery, Cleveland Clinic, Ohio will perform the procedures with 2D and 3D laparoscopy. Each surgeon will perform 9 total colectomies with 3D, and 9 total colectomies with the 2D laparoscopy system. In total, 54 patients will be included (27 patients for each group).

ELIGIBILITY:
Inclusion Criteria:

* Indication for surgery must be Ulcerative Colitis
* Patient age between 18 and 80
* Elective procedure
* BMI between 17 and 30
* Total colectomy with end ileostomy, without proctectomy

Exclusion Criteria:

* Any preoperative diagnosis other than UC
* Patient age< 18, or >80
* Emergency surgery
* Previous gastrointestinal surgery
* BMI>30
* Pregnancy
* Presence of any gastrointestinal tract malignancy
* Segmental colon resections, completion proctectomy, total proctocolectomy, pouch procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-03; Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emre Gorgun, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 3D Visualization: 3-dimensional visualization: In this group, total laparoscopic abdominal colectomy will be performed for patients diagnosed with ulcerative colitis by using 3D Laparoscopic Surgical Video System.
  This group will be consisted of 27 patients, 9 colectomies performed by 3 surgeons.Effect of using 3D Laparoscopic Surgical Video System on operative outcomes will be evaluated.
  3-dimensional visualization: Subjects are receiving Standard of Care Colectomy for Ulcerative Colitis visualized in 3D mode
- 2D Visualization: 2-dimensional visualization: In this group, total laparoscopic abdominal colectomy will be performed for patients diagnosed with ulcerative colitis by using conventional Laparoscopic Surgical Video System.
  This group will be consisted of 27 patients, 9 colectomies performed by 3 surgeons and outcomes will be evaluated.
  2-dimensional visualization: Subjects are receiving Standard of Care Colectomy for Ulcerative Colitis visualized in 2D mode
Period: Overall Study
Arm/Group | 3D Visualization | 2D Visualization
Started | 27 | 26
Completed | 27 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3D Visualization | 2D Visualization | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 21 | 46
  >=65 years | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 53 subjects total were included in analysis
  years | 36.8 (15.2) | 43.2 (17.0) | 40.0 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 16 | 14 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 53
Average BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.0 (4.25) | 23.9 (5.17) | 23.5 (4.72)

OUTCOME MEASURES:

1. Primary Outcome: Operating Time
Description: total operating time
Time Frame: 180 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 3D Visualization | 2D Visualization
Number analyzed (Participants) | 27 | 26
minutes | 75.3 (30.8) | 82.7 (38.6)

2. Secondary Outcome: Major Complication
Description: Number of Participants with Intraoperative Complications
Time Frame: 180 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 3D Visualization | 2D Visualization
Number analyzed (Participants) | 27 | 26
Participants | 8 | 8

ADVERSE EVENTS:
Time Frame: The standard post-operative period of 30 days.
Arm/Group | 3D Visualization | 2D Visualization
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 8/27 | 7/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3D Visualization (N=27) | 2D Visualization (N=26)
Post-operative ileus (Surgical and medical procedures) | 4 (4) | 1 (1)
Wound Dehiscence (Surgical and medical procedures) | 1 (1) | 0 (0)
Portal vein thrombosis/Deep vein thrombosis (Surgical and medical procedures) | 0 (0) | 2 (2)
Surgical Site Infection (Surgical and medical procedures) | 0 (0) | 2 (2)
Readmission (Surgical and medical procedures) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT02370056/Prot_SAP_001.pdf
  • Informed Consent Form (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT02370056/ICF_000.pdf